CLINICAL TRIAL: NCT01128556
Title: The Evaluation of the Effect of Bepreve, a Topical Ocular Antihistamine, on the Measurement of Wheal and Flare Response From Histamine Skin Prick Testing
Brief Title: The Evaluation of Bepreve on the Measurement of Wheal and Flare Response From Histamine Skin Prick Testing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: North Texas Institute for Clinical Trials (Other)
Responsible Party: Bob Q. Lanier, M.D., North Texas Institute for Clinical Trials
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: MAC-01-10
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2010-07

CONDITIONS: Histamine Responsive Allergy Patients
Keywords: allergic conjunctivitis; histamine skin testing
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — bepotastine besilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bepreve (Experimental): topical ocular treatment as indicated
  Interventions: Drug: Bepreve; Drug: Refresh Tears

INTERVENTIONS:
Drug: Bepreve — Bepreve (bepotastine besilate ophthalmic solution 1.5%) one drop in each eye twice daily
  Other Names: bepotastine besilate
Drug: Refresh Tears — Refresh Tears one drop to each eye twice daily for 7 days after the conclusion of Bepreve treatment

SUMMARY:
To evaluate the effect of BEPREVE compared to a REFRESH Tears Lubricant eye drop on the measurement of the wheal and flare from histamine skin prick testing. This is an open label, two-week, post-marketing study conducted on histamine responsive patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, 18 to 65 years of age
* Patients must demonstrate a positive reaction to a Histamine skin-prick test. Manifested by a histamine-induced wheal of >3mm in diameter over the normal saline control after 15 minutes of elapsed time

Exclusion Criteria:

* Significant signs and symptoms of currently active allergic disease (SAR, perennial allergic rhinitis, episodic allergic rhinitis)
* Upper respiratory tract infection, sinusitis, asthma or flu-like symptoms within 2 weeks prior to visit 1
* Subjects who have dermatographism or other skin conditions which might interfere with the interpretation of the skin test results
* Subjects who are receiving escalating doses of immunotherapy, oral immunotherapy or short course (rush) immunotherapy
* Known hypersensitivity to the investigational product or to drugs with similar chemical properties
* Pregnancy and/or breast feeding
* Use of antihistamines, NSAIDS, steroids, or other drugs which may affect the skin-response
* Use of any medications or agents that are not specified above that may confound the interpretation of the results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
measurement of Wheal and Flare response from histamine skin-prick testing | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Bob Q Lanier, MD, Principal Investigator — North Texas Institute for Clinical Trials
Locations (1):
- North Texas Institute for Clinical Trials, Fort Worth, Texas, United States